CLINICAL TRIAL: NCT00526370
Title: Expression of Oncogenic Human Papillomavirus E6/E7 Protein in Tampon Self-Tests
Status: Completed | Type: Observational
Sponsor: University of Aarhus (Other)
Responsible Party: Else Toft Würtz, Student
Other Study IDs: TP07-2351
Record Dates: First submitted 2007-09-06; First posted 2007-09-10 (Estimated); Last update posted 2008-08-13 (Estimated); Status verified 2008-08

CONDITIONS: Normal Uterine Cervical Cytology; Uterine Cervical Dysplasia; Uterine Cervical Neoplasms
Keywords: self test; PAP smear; tampon test; E6/E7; mRNA; HPV
MeSH Terms: conditions — Uterine Cervical Dysplasia; Uterine Cervical Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Tampon self-test from cervix
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- A: Women with at least moderate dysplasia in biopsies from cervix uteri
- B: Women with only normal PAP-smears

SUMMARY:
The purpose of this study is to examine for HPV E6/E7 mRNA in tampon self-tests, and compare with the cytological and histological diagnoses.

Study Hypothesis: Expression of HPV E6/E7 mRNA in Tampon self-tests are a suitable alternative to the routine cervical smear.

ELIGIBILITY:
Inclusion Criteria:

* Women with cervical dysplasia been referred to conisation.
* Women invited to cervical screening program and with only normal smear and normal smears in their history.

Exclusion Criteria:

* Women not performing the tampon self-test before conisation.
* Women not performing the tampon self-test at least 3 month after having a normal PAP-smear taken.

Min Age: 23 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 50 women in out-patient gynecological ward in account of cervical cell changes and 50 women in the national screening program for cervical cancer, included by their G.P.
Sampling Method: Non-Probability Sample
Enrollment: 72 (Actual)
Dates: Start 2007-08; Primary Completion 2008-02 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
Sensitivity and specificity of the HPV test of the material from the tampon self-test | Spring 2008

CONTACTS AND LOCATIONS:
Overall Officials: Hans Svanholm, Head of department, Study Director — Region Hospital, Department of Pathology
Locations (1):
- Region Hospital Randers, Randers, Denmark